CLINICAL TRIAL: NCT02555878
Title: Efficacy and Safety of Rivaroxaban Prophylaxis Compared With Placebo in Ambulatory Cancer Patients Initiating Systemic Cancer Therapy and at High Risk for Venous Thromboembolism
Brief Title: A Study to Evaluate the Efficacy and Safety of Rivaroxaban Venous Thromboembolism (VTE) Prophylaxis in Ambulatory Cancer Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR107047; 39039039STM4001 (Other: Janssen Research & Development, LLC); 2015-001630-21 (EudraCT Number)
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Neoplasms
Keywords: Cancer; Rivaroxaban; Venous thromboembolism
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Participants will be administered rivaroxaban 10 milligram (mg) tablet orally once daily for 180 days.
  Interventions: Drug: Rivaroxaban
- Placebo (Experimental): Participants will be administered matching placebo tablet orally once daily for 180 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 10 milligram (mg) tablet will be administered orally once daily for 180 days.
  Arms: Rivaroxaban
Drug: Placebo — Placebo tablet will be administered orally once daily for 180 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that rivaroxaban is superior to placebo for reducing the risk of the primary composite outcome as defined by objectively confirmed symptomatic lower extremity proximal deep vein thrombosis (DVT), asymptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, symptomatic non-fatal pulmonary embolism (PE), incidental PE, and venous thromboembolism (VTE)-related death in ambulatory adult participants with various cancer types receiving systemic cancer therapy who are at high risk of developing a VTE.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, superiority study comparing the efficacy and safety of rivaroxaban with placebo for primary prophylaxis of venous thromboembolism (VTE) in ambulatory adult participants, with various cancer types who are scheduled to initiate systemic cancer therapy. The study consists of 3 Phases: Screening Phase (14 Days), double-blind treatment Phase (180 Days) and follow up Phase (30 Days). The duration of participation in the study for each participant is approximately 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed solid malignancy including but not limited to: pancreas, lung, stomach, colon, rectum, bladder, breast, ovary, renal or lymphoma (hematologic), with locally advanced or metastatic disease
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Have a Khorana thromboembolic risk Score greater than or equal to (>=) 2
* Creatinine clearance (CrCl) >= 30 milliliter per minute (mL/min)
* Plan to initiate systemic cancer therapy within plus or minus (+-) 1 week of receiving the first dose of study drug with the intention of receiving systemic cancer therapy during the double-blind treatment period for an intended duration determined by the treating oncologist according to standard protocols of clinical care

Exclusion Criteria:

* Diagnosis of primary brain tumors
* Known history of brain metastases
* Bleeding diathesis, hemorrhagic lesions, active bleeding, and other conditions with a high risk for bleeding
* Hematologic malignancies with the exception of lymphoma
* Platelet count less than (<) 50,000/millimeter^3 (mm^3), Life expectancy of less than or equal to (<=) 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (151):
- United States (70):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Martinez, California
  - Santa Barbara, California
  - Torrance, California
  - Upland, California
  - Denver, Colorado
  - Norwich, Connecticut
  - Gainesville, Florida
  - Miami, Florida
  - Miami Shores, Florida
  - New Port Richey, Florida
  - Atlanta, Georgia
  - Evanston, Illinois
  - Joliet, Illinois
  - Peoria, Illinois
  - Rockford, Illinois
  - Skokie, Illinois
  - Urbana, Illinois
  - Anderson, Indiana
  - Cedar Rapids, Iowa
  - Brewer, Maine
  - Baltimore, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Kansas City, Missouri
  - Grand Island, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Albany, New York
  - East Syracuse, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Cleveland, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Erie, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - North Charleston, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Denton, Texas
  - Flower Mound, Texas
  - Garland, Texas
  - Houston, Texas
  - Paris, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Temple, Texas
  - The Woodlands, Texas
  - Tyler, Texas
  - Waco, Texas
  - Roanoke, Virginia
  - Winchester, Virginia
  - Green Bay, Wisconsin
  - Weston, Wisconsin
- Belgium (7):
  - Amberloup
  - Bonheiden
  - Brussels
  - Edegem
  - Laken (brussel)
  - Turnhout
  - Wilrijk
- Brazil (14):
  - Barretos
  - Caxias do Sul
  - Curitiba
  - Itajaí
  - Lajeado
  - Londrina
  - Mogi das Cruzes
  - Porto Alegre
  - Porto Alegre, Rs
  - Rio de Janeiro
  - Santo André
  - São José do Rio Preto
  - São Paulo
  - Sorocaba
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Canada (3):
  - Toronto, Ontario
  - Saint-Jérôme, Quebec
  - Québec
- Czechia (10):
  - Benešov nad Černou
  - Brno
  - Jindřichův Hradec
  - Kladno
  - Liberec
  - Nový Jičín
  - Olomouc
  - Pardubice
  - Prague
  - Tábor
- France (9):
  - Angers
  - Avignon
  - Dijon
  - Hyers
  - Le Mans
  - Paris
  - Rennes
  - Saint-Herblain
  - Valenciennes
- Germany (20):
  - Berlin
  - Brandenburg
  - Cologne
  - Dortmund
  - Dresden
  - Esslingen am Neckar
  - Gauting
  - Hamburg
  - Hanover
  - Herne
  - Kiel
  - Leipzig
  - Lübeck
  - Magdeburg
  - Merseburg
  - Minden
  - München
  - Paderborn
  - Recklinghausen
  - Weiden
- Russia (9):
  - Arkhangelsk
  - Chelyabinsk
  - Kursk
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Tomsk
  - Yaroslavi
- United Kingdom (7):
  - Bournemouth
  - Cheltenham
  - Dundee
  - London
  - Manchester
  - Plymouth
  - Swindon

REFERENCES:
- [Derived] Khorana AA, Barnard J, Wun T, Vijapurkar U, Damaraju CV, Moore KT, Wildgoose P, McCrae KR. Biomarker signatures in cancer patients with and without venous thromboembolism events: a substudy of CASSINI. Blood Adv. 2022 Feb 22;6(4):1212-1221. doi: 10.1182/bloodadvances.2021005710. PMID 34807979
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Vadhan-Raj S, McNamara MG, Venerito M, Riess H, O'Reilly EM, Overman MJ, Zhou X, Vijapurkar U, Kaul S, Wildgoose P, Khorana AA. Rivaroxaban thromboprophylaxis in ambulatory patients with pancreatic cancer: Results from a pre-specified subgroup analysis of the randomized CASSINI study. Cancer Med. 2020 Sep;9(17):6196-6204. doi: 10.1002/cam4.3269. Epub 2020 Jul 14. PMID 32663379
- [Derived] Khorana AA, Soff GA, Kakkar AK, Vadhan-Raj S, Riess H, Wun T, Streiff MB, Garcia DA, Liebman HA, Belani CP, O'Reilly EM, Patel JN, Yimer HA, Wildgoose P, Burton P, Vijapurkar U, Kaul S, Eikelboom J, McBane R, Bauer KA, Kuderer NM, Lyman GH; CASSINI Investigators. Rivaroxaban for Thromboprophylaxis in High-Risk Ambulatory Patients with Cancer. N Engl J Med. 2019 Feb 21;380(8):720-728. doi: 10.1056/NEJMoa1814630. PMID 30786186
- [Derived] Khorana AA, Vadhan-Raj S, Kuderer NM, Wun T, Liebman H, Soff G, Belani C, O'Reilly EM, McBane R, Eikelboom J, Damaraju CV, Beyers K, Dietrich F, Kakkar AK, Riess H, Peixoto RD, Lyman GH. Rivaroxaban for Preventing Venous Thromboembolism in High-Risk Ambulatory Patients with Cancer: Rationale and Design of the CASSINI Trial. Rationale and Design of the CASSINI Trial. Thromb Haemost. 2017 Nov 1;117(11):2135-2145. doi: 10.1160/TH17-03-0171. Epub 2017 Sep 21. PMID 28933799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 841 participants were enrolled in the study to receive either of the 2 treatments: rivaroxaban or matching placebo.
Pre-assignment Details: Deaths which were primary cause of treatment discontinuation (up to Day 180) are reported in participant flow excluding deaths which occurred after discontinuation.
Groups:
- Placebo: Participants received placebo tablet matched to rivaroxaban orally once daily for 180 days.
- Rivaroxaban 10 mg: Participants received rivaroxaban 10 milligram (mg) tablet orally once daily for 180 days.
Period: Overall Study
Arm/Group | Placebo | Rivaroxaban 10 mg
Started | 421 | 420
Treated | 404 | 405
Completed | 255 | 270
Not Completed | 166 | 150
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 48 | 48
Not completed — Adverse Event | 12 | 8
Not completed — Death | 74 | 59
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 12 | 13
Not completed — Other | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rivaroxaban 10 mg | Total
Number analyzed (Participants) | 421 | 420 | 841
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.19) | 62.1 (11.22) | 62 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 198 | 413
  Male | 206 | 222 | 428
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 63 | 132
  Not Hispanic or Latino | 312 | 314 | 626
  Unknown or Not Reported | 40 | 43 | 83
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  White | 346 | 352 | 698
  Black | 18 | 13 | 31
  Asian | 5 | 6 | 11
  Other | 21 | 10 | 31
  Not reported | 31 | 39 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 3 | 10 | 13
  Brazil | 55 | 48 | 103
  Bulgaria | 15 | 19 | 34
  Canada | 0 | 3 | 3
  Czech Republic | 25 | 12 | 37
  France | 29 | 34 | 63
  Germany | 60 | 53 | 113
  Italy | 17 | 15 | 32
  Russian Federation | 59 | 61 | 120
  United Kingdom | 30 | 19 | 49
  United States of America | 128 | 146 | 274

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Time to First Occurrence of Primary Efficacy Endpoint (Composite and Components)
Description: Percentage of participants with time to the first occurrence of primary efficacy endpoint (composite and components) was reported. The primary efficacy composite endpoint is time to first occurrence of objectively confirmed symptomatic and asymptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, symptomatic non-fatal PE, incidental PE, or VTE-related death as adjudicated by an independent blinded Clinical Endpoint Committee (CEC).
Time Frame: Up to Day 180
Population: The Intent-to-treat (ITT) population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants
  Primary efficacy composite endpoint | 8.79 | 5.95
  Symptomatic lower extremity proximal DVT | 1.90 | 2.14
  Symptomatic lower extremity distal DVT | 1.19 | 0.48
  Symptomatic upper extremity DVT | 1.43 | 0.95
  Symptomatic non-fatal PE | 1.19 | 1.19
  Asymptomatic lower extremity proximal DVT | 2.61 | 0.95
  Incidental PE | 2.38 | 1.43
  VTE-related death | 0.71 | 0.24
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for primary efficacy composite endpoint; Test type: Superiority; p = 0.101, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.40 to 1.09]
Statistical Analysis 2: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for Symptomatic lower extremity proximal DVT; Test type: Superiority; p = 0.814, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.43 to 2.91]
Statistical Analysis 3: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for symptomatic lower extremity distal DVT; Test type: Superiority; p = 0.260, Log Rank; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.08 to 2.07]
Statistical Analysis 4: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for symptomatic upper extremity DVT; Test type: Superiority; p = 0.538, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.19 to 2.39]
Statistical Analysis 5: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for symptomatic non-fatal PE; Test type: Superiority; p = 0.977, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.29 to 3.52]
Statistical Analysis 6: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for asymptomatic lower extremity proximal DVT; Test type: Superiority; p = 0.063, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.11 to 1.11]
Statistical Analysis 7: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for incidental PE; Test type: Superiority; p = 0.301, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.21 to 1.62]
Statistical Analysis 8: Comparison: Placebo vs Rivaroxaban 10 mg; Statistical analysis for VTE-related death; Test type: Superiority; p = 0.314, Log Rank; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.03 to 3.18]

2. Primary Outcome: Percentage of Participants With Time to the First Occurrence of Major Bleeding Events as Defined by International Society of Thrombosis and Haemostasis (ISTH)
Description: Major bleeding is defined as clinically overt bleeding that is associated with a reduction in hemoglobin of 2 gram per deciliter (g/dL) or more, or a transfusion of 2 or more units of packed red blood cells or whole blood, or occurrence at a critical site defined as intracranial, intra-spinal, intraocular, pericardial, intra-articular, intra-muscular with compartment syndrome, retroperitoneal, or fatal outcome.
Time Frame: From first dose of study drug to 2 days after the last dose of the study drug (up to 32 weeks)
Population: The safety analysis population consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 404 | 405
Percentage of participants | 0.99 | 1.98
Statistical Analysis 1: Comparison: Placebo vs Rivaroxaban 10 mg; Test type: Superiority; p = 0.265, Log Rank; Hazard Ratio (HR) = 1.96, 95% CI 2-sided [0.59 to 6.49]

3. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Symptomatic VTE Events or VTE-Related Deaths
Description: Percentage of participants with time to first occurrence of the composite endpoint of symptomatic VTE events (symptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, or symptomatic non-fatal PE) or VTE related deaths as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 5.23 | 3.81

4. Secondary Outcome: Percentage of Participants With All-Cause Mortality
Description: Percentage of participants with all-cause mortality as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported. Overall deaths occurred during observation period (defined by start to end date of the observation period [that is approximately 180 days] are reported here.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 23.8 | 20.0

5. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Fatal or Non-fatal Arterial Thromboembolic Events (ATE)
Description: Percentage of participants with time to first occurrence of fatal/non-fatal ATE (a composite of occurrence of myocardial infarction (MI), stroke [ischemic infarction with or without hemorrhagic conversion or primary hemorrhagic events - intraparenchymal hemorrhage, subdural hematoma or epidural hematoma] or any other ATE recorded) event as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 1.66 | 0.95

6. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Fatal or Non-fatal Visceral VTE
Description: Percentage of participants with time to the first occurrence of fatal or non-fatal visceral VTE as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 0.48 | 0.24

7. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Composite Efficacy Endpoint 1
Description: Percentage of participants with time to first occurrence of composite efficacy endpoint 1 (composite of objectively confirmed symptomatic and asymptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, symptomatic non-fatal PE, incidental PE or all-cause mortality) as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 29.5 | 23.1

8. Secondary Outcome: Percentage of Participants With Time to First Occurrence of Composite Efficacy Endpoint 2
Description: Percentage of participants with time to first occurrence of composite efficacy endpoint 2 (composite of objectively confirmed symptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, symptomatic non-fatal PE or VTE-related deaths) as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 5.23 | 3.81

9. Secondary Outcome: Percentage of Participants With Time to First Occurrence of Composite Efficacy Endpoint 3
Description: Percentage of participants with time to first occurrence of composite efficacy endpoint 3 (composite of objectively confirmed symptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, asymptomatic lower extremity proximal DVT, symptomatic non-fatal PE, incidental PE, VTE-related deaths, fatal/non-fatal ATE [MI, stroke {ischemic infarction with or without hemorrhagic conversion or primary hemorrhagic events - intraparenchymal hemorrhage, subdural hematoma or epidural hematoma} or any ATE] or fatal/non-fatal visceral VTE) as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 10.7 | 6.90

10. Secondary Outcome: Percentage of Participants With Time to First Occurrence of Composite Efficacy Endpoint 4
Description: Percentage of participants with time to first occurrence of composite efficacy endpoint 4 (composite of objectively confirmed symptomatic lower extremity proximal DVT, symptomatic lower extremity distal DVT, symptomatic upper extremity DVT, symptomatic non-fatal PE, VTE-related deaths or major bleeding events up to Day 180) as adjudicated by an independent blinded CEC up-to-Day 180 observation period was reported.
Time Frame: Up to Day 180
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 421 | 420
Percentage of participants | 6.89 | 5.71

11. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Clinically Relevant Non-major Bleeding
Description: Percentage of participants with time to the first occurrence of clinically relevant non-major bleeding was reported. Clinically relevant non-major bleeding is defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, or unscheduled contact with a physician, or temporary cessation of study treatment, or discomfort such as pain, or impairment of activities of daily life.
Time Frame: From first dose of study drug to 2 days after the last dose of the study drug (up to 32 weeks)
Population: The safety analysis population consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 404 | 405
Percentage of participants | 1.98 | 2.72

12. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Minor Bleeding
Description: Percentage of participants with time to the first occurrence of minor bleeding was reported. Minor bleeding (that is, minimal bleeding) is defined as overt bleeding episodes not meeting the criteria for major or clinically relevant non-major bleeding event.
Time Frame: From first dose of study drug to 2 days after the last dose of the study drug (up to 32 weeks)
Population: The safety analysis population consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 404 | 405
Percentage of participants | 3.96 | 6.91

13. Secondary Outcome: Percentage of Participants With Time to the First Occurrence of Any Bleeding
Description: Percentage of participants with time to the first occurrence of any bleeding event was reported. Any bleeding is defined as a composite of major bleeding, clinically relevant non-major bleeding, or minor bleeding.
Time Frame: From first dose of study drug to 2 days after the last dose of the study drug (up to 32 weeks)
Population: The safety analysis population consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rivaroxaban 10 mg
Number analyzed (Participants) | 404 | 405
Percentage of participants | 6.44 | 11.1

ADVERSE EVENTS:
Time Frame: Up to 32 weeks
Description: The safety analysis population consisted of all randomized participants who received at least 1 dose of study drug. Deaths occurred throughout the study are reported below.
Arm/Group | Placebo | Rivaroxaban 10 mg
All-Cause Mortality (participants affected / at risk) | 106/404 | 85/405
Serious Adverse Events (participants affected / at risk) | 128/404 | 134/405
Other Adverse Events (participants affected / at risk) | 145/404 | 138/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=404) | Rivaroxaban 10 mg (N=405)
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Cardiotoxicity (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 | 1
Intestinal Infarction (Gastrointestinal disorders) | 0 | 1
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Chest Pain (General disorders) | 1 | 0
Condition Aggravated (General disorders) | 0 | 1
Death (General disorders) | 2 | 0
Disease Progression (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 4 | 5
Generalised Oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Mucosal Inflammation (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 8
Bile Duct Obstruction (Hepatobiliary disorders) | 3 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal Sepsis (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Atypical Pneumonia (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Biliary Sepsis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 3
Cholecystitis Infective (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 1
Febrile Infection (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Klebsiella Sepsis (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 0
Lung Infection (Infections and infestations) | 1 | 2
Neutropenic Sepsis (Infections and infestations) | 3 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 10
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 6
Septic Shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 3
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 1
Aspiration Bronchial (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 2
General Physical Condition Abnormal (Investigations) | 0 | 1
Glomerular Filtration Rate Decreased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Feeding Intolerance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 | 29
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Muscle Contractions Involuntary (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient Global Amnesia (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 3
Dysuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=404) | Rivaroxaban 10 mg (N=405)
Anaemia (Blood and lymphatic system disorders) | 59 | 46
Neutropenia (Blood and lymphatic system disorders) | 24 | 25
Constipation (Gastrointestinal disorders) | 12 | 29
Diarrhoea (Gastrointestinal disorders) | 36 | 34
Nausea (Gastrointestinal disorders) | 55 | 55
Vomiting (Gastrointestinal disorders) | 17 | 28
Fatigue (General disorders) | 32 | 44
Decreased Appetite (Metabolism and nutrition disorders) | 25 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT02555878/SAP_000.pdf
  • Study Protocol (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT02555878/Prot_001.pdf